CLINICAL TRIAL: NCT04373226
Title: Study of Arithmetic Abilities of Children With 22q11.2 Deletion Syndrome Aged From 4 to 11 Years Old
Brief Title: Arithmetic Abilities in Children With 22q11.2DS
Acronym: ARITH22
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Departure of the investigator who was recruiting subjects
Sponsor: Hôpital le Vinatier (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2020-A00102-37
Record Dates: First submitted 2020-04-30; First posted 2020-05-04 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: 22q11.2 Deletion Syndrome
Keywords: 22q11.2 deletion syndrome; arithmetic; magnitude representation; children
MeSH Terms: conditions — DiGeorge Syndrome | interventions — Neuropsychological Tests

STUDY DESIGN:
Intervention Model Description: Monocentric study with two parallel groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 22q11.2DS (Experimental): Children aged from 4 to 11 years old with 22q11.2 deletion syndrome
  Interventions: Behavioral: Magnitude comparison tasks and neuropsychological testing
- NON22q11.2DS (Active Comparator): Children aged from 4 to 11 years old without developmental disease
  Interventions: Behavioral: Magnitude comparison tasks and neuropsychological testing

INTERVENTIONS:
Behavioral: Magnitude comparison tasks and neuropsychological testing — neuropsychological testing (ZAREKI-R) and magnitude comparison tasks with stimuli of different types (visual, visuo-spatial)

SUMMARY:
The study ARITH22 will investigate the role of visuo-spatial attention on arithmetic abilities of children with 22q11.2 deletion syndrome.

DETAILED DESCRIPTION:
Children with 22q11.2 deletion syndrome often have arithmetic learning disability because of magnitude representation impairment. Previous works suggested that magnitude representation impairment could be a result of endogenous visuo-spatial attention dysfunction in 22q11.2DS. Nevertheless this relationship is still poor explored. The influence of visuo-spatial abilities on arithmetic achievement could also be modulated by developmental age. The study ARITH22 will test these hypotheses thanks to magnitude comparisons tasks, in children with 22q11.2 deletion syndrome and matched children without developmental disease.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of 22q11.2 deletion syndrome or no developmental disease
* Aged from 4 to 11 years old
* French language

Exclusion Criteria:

* Diagnosis of intellectual deficiency according to DSM 5 criteria
* Drug prescribed for somatic condition that could influence cerebral functioning

Ages: 4 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 41 (Actual)
Dates: Start 2020-09-16 (Actual); Primary Completion 2023-04-14 (Actual); Study Completion 2023-04-14 (Actual)

PRIMARY OUTCOMES:
Percentage of impaired scaled score | single day
  percentage of impaired scaled score at ZAREKI-R

SECONDARY OUTCOMES:
Percentage of correct responses | single day
  percentage of correct responses in magnitude comparisons tasks
Mean reaction time | single day
  mean reaction time in magnitude comparison tasks

CONTACTS AND LOCATIONS:
Overall Officials: Caroline DEMILY, MD PH, Principal Investigator — Centre Hospitalier le Vinatier
Locations (1):
- Hopital Vinatier, Lyon, Auvergne-Rhône-Alpes, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Favre E, Piveteau M, Babinet MN, Demily C. Extent of magnitude representation deficit and relationship with arithmetic skills in children with 22q11.2DS. Orphanet J Rare Dis. 2024 Jul 3;19(1):250. doi: 10.1186/s13023-024-03263-1. PMID 38961462